CLINICAL TRIAL: NCT05361109
Title: An Open-Label Pilot Study to Evaluate the Efficacy and Safety of Baricitinib in Subjects With Cutaneous Dermatomyositis
Brief Title: Baricitinib for Cutaneous Dermatomyositis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty recruiting subjects
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Kwanghoon (Bobby) Han, Clinical Associate Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00014444; CUDM001 (Other: Principal Investigator)
Record Dates: First submitted 2022-04-03; First posted 2022-05-04 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Dermatomyositis
Keywords: cutaneous; dermatomyositis; baricitinib
MeSH Terms: conditions — Dermatomyositis | interventions — baricitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Barcitinib (Experimental): All subjects will initially receive baricitinib 2mg daily for 8 weeks. If no unexpected serious adverse events related to baricitinib have occurred during the first 8 weeks of treatment in the opinion of the investigator, the dose will be increased to 4 mg daily for 16 weeks.
  Interventions: Drug: Baricitinib

INTERVENTIONS:
Drug: Baricitinib — The investigational medicinal product (IP) for this study is baricitinib 2mg. The dose will be administered as one 2mg tablet by mouth once daily for the first 8 weeks of study. If no unexpected serious adverse events related to baricitinib in the opinion of the investigator occur during the first 8 weeks of treatment, the dose will be increased to two 2mg tablets (4mg daily) for the remaining 16 weeks of study. All study participants will take baricitinib in combination with standard of care background therapy.
  Other Names: Olumiant

SUMMARY:
This is a phase 2, single-center study in patients with active cutaneous DM who have had an inadequate response. An inadequate response is defined as no improvement with standard of care treatment based on the investigator's opinion.

All subjects will initially receive baricitinib 2mg daily for 8 weeks. If no unexpected serious adverse events related to baricitinib have occurred during the first 8 weeks of treatment in the opinion of the investigator, the dose will be increased to 4 mg daily for 16 weeks. Visits are scheduled at baseline, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks, and 24 weeks. Evaluation of primary endpoint occurs at week 24. All subjects receive a phone call from study

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-nursing female
2. Age ≥18 years at time of consent
3. Typical cutaneous DM manifestations including heliotrope rash, Gottron's papules/sign, V-sign, shawl sign, holster sign, confirmed by skin biopsy, with or without DM muscle disease classified based on the Bohan and Peter criteria at screening and baseline visit
4. Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI) activity score ≥ 12 corresponding to moderate to severe disease activity at screening and baseline visit
5. Active disease (i.e., CDASI ≥ 12) despite adequate prior treatment experience with corticosteroids, immunosuppressants, or biologics
6. Patients taking methotrexate must be on a stable dose for at least 4 weeks prior to baricitinib initiation
7. Patients who have received mycophenolate, azathioprine, cyclosporine, or tacrolimus must have discontinued for at least 4 weeks prior to signing the informed consent.
8. Patients who have received IVIG, rituximab or any other biologic agents must have discontinued for at least 6 months prior to signing the informed consent
9. Patients taking oral corticosteroids, the dose must be ≤ 15 mg/day prednisone or equivalent and not be changed for 2 weeks prior to baseline visit
10. Females of childbearing potential and males with female partners of childbearing potential may participate in this study only if using a highly effective method of contraception

Highly Effective Methods of Contraception:

1. A tubal ligation, or surgical sterilization
2. FDA approved hormonal contraceptive such as oral contraceptives, emergency contraception used as directed, patches, implants, injections, rings, or hormonally impregnated intrauterine device (IUD)
3. Intrauterine device (IUD)
4. Abstinence if this method of contraception coincides with normal lifestyle choice of the participant. Abstinence for the duration of the study is not an acceptable method of contraception for the purposes of this study.

Exclusion Criteria:

1. Previous treatment with baricitinib.
2. Previous treatment with tofacitinib or updacitinib.
3. Current use of strong Organic Anion Transporters 3 (OAT3) inhibitors including probenecid.
4. Uncontrolled or rapidly progressive myositis or interstitial lung disease at the discretion of the investigator which is likely to warrant escalation in therapy beyond permitted background medications.
5. Cancer-associated myositis (myositis diagnosed within 2 years of a diagnosis of cancer).
6. Patients who are known to be positive for the anti-TIF1-γ (p155/140) or anti-NXP2 autoantibody unless they are determined not to be associated with malignancy at the discretion of the investigator.
7. Other inflammatory diseases that might confound the evaluations of efficacy including but not limited to rheumatoid arthritis (RA), systemic lupus erythematosus (SLE), psoriatic arthritis, inflammatory bowel disease.
8. Recurrent or chronic bacterial, viral, fungal, mycobacterial, or other infections including HIV, Hepatitis B or C, latent TB (TB not adequately treated according to guidelines)
9. History of recurrent herpes zoster, disseminated (multi-dermatomal) herpes zoster, disseminated herpes simplex or ophthalmic zoster. Herpes zoster lesions within 90 days prior to screening.
10. Primary or secondary immunodeficiency.
11. Current uncontrolled renal, gastrointestinal, endocrine, pulmonary, cardiac, or neurologic disease, which, in the opinion of the investigator, might place the patient at unacceptable risk for participation in this study.
12. History of malignancy within 5 years prior to screening, except for appropriately treated carcinoma in situ of the cervix and non-melanoma skin carcinoma.
13. History of lymphoproliferative disease, including lymphoma, and monoclonal gammopathy of undetermined significance.
14. History of venous thromboembolism, including deep vein thrombosis and pulmonary embolism.
15. History of alcohol, drug, or chemical abuse within one year prior to signing the informed consent form.
16. Laboratory exclusion criteria within 60 days of Consent including

    * Hemoglobin (Hgb) < 8g/dL
    * White Blood Count (WBC) < 3,000/μL fidential Page 13 of 40
    * Absolute Neutrophil Count (ANC) < 1,500/μL
    * Absolute Lymphocyte Count (ALC) < 800/μL
    * Platelets < 100,000/μL
    * eGFR < 60 ml/min
    * ALT or AST >1.5 times ULN not due to DM.
17. Major surgery within 8 weeks prior to Screening or planned major surgery at any time during participation in the study.
18. Immunization with a live/attenuated vaccine within 4 weeks prior to Screening.
19. Pregnant or nursing women, or women of child-bearing potential who plan to become pregnant prior to 14 weeks after the last dose of baricitinib treatment.
20. Patients of reproductive potential not willing to use a highly effective method of contraception as defined in Section 5.3.1.10.
21. Prisoners, or subjects who are compulsory detained, or cannot provide informed consent without the use of a legally authorized representative (LAR).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Cutaneous Disease Activity Severity Index (CDASI) activity score | 24 Weeks
  Change in Cutaneous Disease Activity Severity Index (CDASI) activity score (0-100), higher scores mean a worse outcome

SECONDARY OUTCOMES:
Cutaneous Disease Activity Severity Index (CDASI) activity score | 12 weeks
  Change in Cutaneous Disease Activity Severity Index (CDASI) activity score (0-100), higher scores mean a worse outcome
International Myositis Assessment & Clinical Studies Group (IMACS) Disease Activity Core Set Measures | 12 weeks and 24 weeks
  Change in International Myositis Assessment & Clinical Studies Group (IMACS) Disease Activity Core Set Measures
SF-36 | 12 weeks and 24 weeks
  Change in SF-36
Dermatology Life Quality Index (DLQI) | 12 weeks and 24 weeks
  Change in Dermatology Life Quality Index (DLQI)
Adverse event | 24 weeks
  Adverse event monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Kwanghoon Han, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States